CLINICAL TRIAL: NCT00091416
Title: A Phase I Clinical Trial to Evaluate the Safety of a Multiclade Recombinant Adenoviral Vector HIV-1 Vaccine Administered to Healthy, HIV-1 Uninfected, Adult Participants Who Received DNA Plasmid Vaccine or Placebo in the HVTN 052 Clinical Trial
Brief Title: Safety of and Immune Response to an HIV-1 Vaccine Boost (VRC-HIVADV014-00-VP) in HIV Uninfected Adults Who Participated in HVTN 052
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 057; 10123 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2004-09-08; First posted 2004-09-09 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: VRC-HIVADV014-00-VP

SUMMARY:
The purpose of this study is to test the safety of and immune response to an HIV-1 vaccine, VRC-HIVADV014-00-VP, when given as a vaccine booster to HIV uninfected adults who participated in HVTN 052.

DETAILED DESCRIPTION:
The worldwide HIV epidemic highlights the importance of developing an affordable, globally successful vaccine for HIV prevention. The VRC-HIVADV014-00-VP adenoviral vector vaccine used in this study was developed to stimulate strong virus-specific CD8 cytotoxic T-lymphocyte (CTL) responses thought to be crucial in an effective preventive HIV vaccine. The purpose of this study is to determine the safety and immunogenicity of a VRC-HIVADV014-00-VP vaccine boost given to healthy, HIV uninfected individuals who participated in HVTN 052, which evaluated the VRC-HIVDNA009-00-VP DNA plasmid vaccine. In that study, participants received either 3 injections of vaccine, 2 injections of vaccine and 1 injection of placebo, or 3 injections of placebo over a 2-month period.

This study will last one year. Participants will be randomly assigned to receive vaccine boost or placebo by intramuscular injection. The injections will be given 6 to 9 months after each participant's first HVTN 052 study injection, preferably as close to 6 months after the first HVTN 052 injection as possible. After a screening visit, study visits will occur at enrollment (when the injection will be given), at Week 2, and at Months 1, 3, 6, and 12. Blood collection, physical exam, and medication assessment will occur at every study visit; urine collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in and have completed all 3 study vaccine injections for HVTN 052
* Understanding of vaccination procedure
* Good general health
* HIV uninfected
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (HCV) antibody negative, or negative for HCV PCR if the anti-HCV is positive
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Immunosuppressive medications within 168 days prior to study
* Blood products within 120 days prior to study
* Immunoglobulin within 60 days prior to study
* Live attenuated vaccines within 30 days prior to study
* Investigational research agents within 30 days prior to study
* Medically indicated subunit or killed vaccines within 14 days prior to study
* Allergy shots within 30 days prior to study
* Current anti-tuberculosis prophylaxis or therapy
* Anaphylaxis or other serious adverse reactions to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection
* Unstable asthma (e.g., daily symptoms; use of oral or orally inhaled corticosteroids or other treatments; emergent care, urgent care, hospitalization, or intubation during the past 2 years)
* Diabetes mellitus. A participant with past gestational diabetes is not excluded.
* Thyroid disease, including removal of thyroid and diagnoses requiring medication. A participant not requiring thyroid medication during the last year is not excluded.
* Serious angioedema. A participant who has had an episode of angioedema over 3 years prior to the study, and has not required medications for at least 2 years, is not excluded.
* Uncontrolled hypertension
* Diagnosis of bleeding disorder
* Malignancy, except those with a surgical excision that has a reasonable assurance of sustained cure and/or is unlikely to recur during the period of the study
* Seizure disorder requiring medication within the last 3 years
* Absence of the spleen
* Mental illness that would interfere with compliance with the protocol
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Peiperl, MD, Study Chair — San Francisco Department of Public Health / University of California - San Francisco; Julie McElrath, MD, PhD, Study Chair — Fred Hutchinson Cancer Research Center / University of Washington
Locations (8):
- United States (8):
  - Johns Hopkins Bloomberg School of Public Health,Ctr for Immunization Research,Project SAVE-Baltimore, Baltimore, Maryland
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Gomez-Roman VR, Robert-Guroff M. Adenoviruses as vectors for HIV vaccines. AIDS Rev. 2003 Jul-Sep;5(3):178-85. PMID 14598567
- [Background] McShane H. Prime-boost immunization strategies for infectious diseases. Curr Opin Mol Ther. 2002 Feb;4(1):23-7. PMID 11883691
- [Background] Pinto AR, Fitzgerald JC, Giles-Davis W, Gao GP, Wilson JM, Ertl HC. Induction of CD8+ T cells to an HIV-1 antigen through a prime boost regimen with heterologous E1-deleted adenoviral vaccine carriers. J Immunol. 2003 Dec 15;171(12):6774-9. doi: 10.4049/jimmunol.171.12.6774. PMID 14662882
- [Background] Shiver JW, Emini EA. Recent advances in the development of HIV-1 vaccines using replication-incompetent adenovirus vectors. Annu Rev Med. 2004;55:355-72. doi: 10.1146/annurev.med.55.091902.104344. PMID 14746526
- See also: Click here for more information about the HVTN 052 study — http://clinicaltrials.gov/show/NCT00071851